CLINICAL TRIAL: NCT03841006
Title: Role of MRI Defecography in Diagnosis of Obstructed Defecation Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alshimaa Abdalkreem (Other)
Responsible Party: Sponsor-Investigator, Alshimaa Abdalkreem, Specialist at radiology department Assiut University hospital, Assiut University
Organization: Assiut University (Other)
Other Study IDs: MR defecpgraphy in ODS
Record Dates: First submitted 2019-02-03; First posted 2019-02-15 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: MRI Defecography, ODS

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: symptomatic patient and suspicious to have ODS by history and clinical examination those patient will have MRI defecography
  Interventions: Device: MRI
- asymptomatic group: Asymptomatic group not suspicious to have ODS by history or clinical examination they will undergone MRI defecography
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — dynamic MRI pelvis

SUMMARY:
The aim of the study was to assess the advantages of dynamic magnetic resonance imaging defecography to elucidate the underlying anatomic and pathophysiologic background in obstructed defecation patients to guide physicians in patient management.

DETAILED DESCRIPTION:
Obstructed defecation syndrome (ODS) is a term used to describe the whole complex of mechanical and functional disorders leading to difficult or inadequate rectal emptying. obstructed defecation syndrome has prevalence rate 3.4 % in general population, In obstructed defecation feces do reach the rectum, but rectal emptying is extremely difficult. These patients have a feeling that defecation is blocked. Despite repetitive attempts, complete evacuation of rectal contents is not possible. The patients may also complain of prolonged and unsuccessful straining at stools, feelings of incomplete evacuation, digital removal of feces, and laxative abuse.

Constipation caused by obstructed defecation is of two basic types: functional and mechanical. The functional type includes anismus (pelvic floor dys-synergy), and descending perineal syndrome, whereas the mechanical type includes rectocele, enterocele, internal intussusception and overt rectal prolapse.

All of these conditions represent either a defect of pelvic support or abnormal function of the pelvic floor musculature. The etiology of ODS is controversial. It is presumed that in childbearing women damage to the innervation and soft tissues of the pelvis may occur as a direct consequence of vaginal childbirth. Trauma to the pelvic soft tissues can result in endopelvic fascial and pelvic support defects. Cumulative nerve damage from stretching of pelvic floor due to childbirth and activities that cause chronic and repetitive increases in intra-abdominal pressure such as obesity and chronic cough have been suggested to play a role in the development of symptomatic defects.

Although patients frequently complain of constipation, symptoms such as fruitless straining and incomplete evacuation are rather subjective and unreliable. Nevertheless, an international team of experts included these symptoms in the definition of constipation.This Rome III guidelines, for a patient to be labeled as suffering from functional constipation, which also includes obstructed defecation, following criteria should be present for at least 3 months:

1. Must include two or more of the following:

   1. Straining during at least 25% of defecations,
   2. Lumpy or hard stools in at least 25% of defecations,
   3. Sensation of incomplete evacuation for at least 25% of defecations,
   4. Sensation of ano-rectal obstruction/ blockage for at least 25% of defecations,
   5. Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor),
   6. Fewer than three defecations per week.
2. Loose stools are rarely present without the use of laxatives.
3. Insufficient criteria for irritable bowel syndrome. The same criteria define dys-synergic defecation as inappropriate contraction of the pelvic floor or less than 20% relaxation of basal resting sphincter pressure with adequate propulsive forces during attempted defecation .

On physical examination, the paradoxical contraction of the pelvic floor can be assessed by palpation of the puborectalis muscle while the patient is straining . Perineal descent >3 cm, mucous discharge or mucosal prolapse may also be seen when the patient is asked to strain for stools . However, most clinicians do not rely on palpation and advocate the use of specific tests to diagnose ODS . Electromyography (EMG) of the pelvic floor, the balloon expulsion test (BET), and defecography are the most frequently used tests. Other radiologic methods for the dynamic evaluation of the ODS include magnetic resonance imaging and ultrasonography, each of which has its advantages and limitations.

The development of fast Magnetic Resonance Imaging sequences provides a new alternative to study all pelvic visceral movements in a dynamic fashion. MR defecography has several important advantages over conventional defecography. Its non-ionic nature, multiplanar capacity, dynamic evaluation and good temporal resolution along with its high-resolution soft-tissue contrast makes it an ideal modality in the assessment of ODS patients. Imaging in the mid-sagittal plane allows evaluation of the anal canal, anorectal angle, levator muscle and hiatus and the vaginal disposition as well as their relationship to a consistent electronically designated pubo-coccygeal Line (PCL). Diagnostic parameters for pelvic dys-synergy include an indented impression of the pubococcygeus muscle on the rectum with excessive obtuse anorectal angulation accompanied by very prolonged rectal emptying on T2-weighted MR images.

ELIGIBILITY:
Inclusion Criteria:

* Patient group: Those with provisional diagnosis of obstructed defecation disorder based on: History by using Rome III criteria. and Physical examination.
* asymptomatic group: will be matched with patients for age and sex.

Exclusion Criteria:

* Any general contraindication of MRI in some cases as presence of paramagnetic substance as pacemakers or in patients with claustrophobia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Assiute university hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
to diagnose obstructed defecation syndrome and its degree by dynamic MRI study with comparison of imaging data with operative data and or clinical scoring of ODS | Baseline
  sensitivity and specificity of MRI defecography in diagnosis of obstructed defecation syndrome and help physician in patient management by using modified Longo score for obstructed defecation syndrome.
  * data collected by history using Rome III guidelines.
  * imaging data :
    1. Normal functional movements of the pelvic floor using pupococygeal line (PCL) as reference line, The anorectal angle (ARA) and Levator plate angle.
    2. Pelvic floor relaxation: using H and M lines
    3. Defecographic disorders: Rectocele, Intussusception, Rectal prolapse ,Descending perineal syndrome, Anismus, or spastic pelvic floor syndrome and Enterocele.
  the imaging data will be correlated with operative data if patient candidate for operation and with clinical examination and modified Longo score patient no candidate for operation.

CONTACTS AND LOCATIONS:
Overall Officials: Gehan Sayed, Study Director — Egypt.Assiut
Locations (1):
- AssiutU university hospital, Asyut, Egypt

REFERENCES:
- [Background] Sakra L, Siller J. [Obstructed defecation syndrome - review article]. Rozhl Chir. 2017 Summer;96(6):247-251. Czech. PMID 28931290